CLINICAL TRIAL: NCT06815783
Title: Reduction of Radiation and Improving Conduction System Pacing Using Ultrasound (CONDUCT USe)
Brief Title: Novel Approach to Conduction System Pacing With Use of Ultrasound
Acronym: CONDUCT USe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Habib Khan (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14539
Record Dates: First submitted 2024-02-21; First posted 2025-02-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Conduction Block, Atrioventricular; Bundle-Branch Block
Keywords: Conduction system pacing; Left bundle branch area pacing; HIS bundle pacing; pacemaker; ultrasound; NTproBNP; EQ5D; LVEF
MeSH Terms: conditions — Atrioventricular Block; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Physicians making the referral for pacing or seeing patients in the future will be masked to whether the patients had ultrasound-guided left bundle branch area pacing. The outcomes assessor will not be aware of whether the patients will be randomized to Group 1 (conventional use of fluoroscopy) or Group 2 (assisted with ultrasound)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Normal deployment of left bundle branch area pacing with use of xrays and fluoroscopy. No use of ultrasound in the procedure.
  Interventions: Device: Fluoroscopy guided
- US guided (Experimental): Patients randomized to this arm will have use of ultrasound in venous access and particularly in attempts to place the pacing lead in the septum at the region of LBBA. This will allow the lead to be directly visualized as it is being passed deep into the septum without perforation and it ensure that the lead is perpendicular to the septum.
  Interventions: Device: Ultrasound guidance

INTERVENTIONS:
Device: Ultrasound guidance — Use of ultrasound in group 2
  Arms: US guided
Device: Fluoroscopy guided — Conventional techniques for implanting LBBAP lead
  Arms: Conventional

SUMMARY:
Each year, over one million pacemakers are implanted globally using x-rays. Recent developments have been aimed at determining which area of the heart is the best option for lead placement. An area in the septum separating the verticals called the left bundle branch area (LBBA) has previously been identified as a safe and effective area for lead placement. However, as the LBBA location is in the center of the heart, it is impossible to see the entire extent using X-ray. Current practice requires x-ray guidance to estimate the location and pacing parameters to confirm proximity. Implanting in LBBA takes longer procedure times and higher exposure to X-ray radiation for both patients and hospital staff. Over time, radiation poses an increased risk of cancer and other medical issues.

This study will determine if using ultrasound can improve pacemaker lead implantation to the LBBA. Benefits to patients may include fewer attempts and more accuracy in lead deployment, thereby reducing risks and providing improved outcomes. Benefits to healthcare delivery may include reduction in total procedure time, thereby allowing more cases per day to reduce waitlist, and reduced X-ray exposure to staff thereby reducing cumulative effects.

ELIGIBILITY:
Inclusion criteria: Patients meeting the following criteria are eligible for the study:

1. Male or female ≥18 years of age
2. Eligible to have a single or dual chamber pacemaker implanted for LBBAP
3. Confirmed diagnosis of conduction tissue disease
4. The participant can understand the written informed consent/assent, provides signed and witnessed written informed consent/assent, and agrees to comply with protocol requirements.
5. Good imaging quality determined on routine echocardiography

Exclusion Criteria: Patients will be excluded if any one of the following criteria is met:

1. Any medical or psychiatric condition that, in the investigator's opinion, could jeopardize or compromise the participant's ability to participate in the study.
2. Any acute active malignancy requiring treatment or life expectancy is deemed less than 1 year.
3. Clinically significant disease that increases their risk of bleeding (hematological disorders, dialysis patient - anticoagulation does not apply)
4. History of alcohol or drug (other than caffeine) use disorder within 12 months of pacemaker implantation.
5. Hepatic impairment defined as ALT/AST >3 × ULN and/or total bilirubin >ULN, at Screening.
6. The participant has any clinically significant illness, in the opinion of the investigator, prior to their pacemaker implantation
7. Any other issues which, in the opinion of the investigator, will make the participant ineligible for study participation.
8. CRT and ICD implants.
9. Pregnancy or female of childbearing age (if negative pregnancy test not provided).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Composite of the Following | During study procedure and through study completion, an average of 12 months
  1. Greater than two attempts at lead deployment to successfully achieve LBBAP
  2. Septal perforation
  3. Worsening tricuspid regurgitation category
  4. Development of LV septal pacing during follow-up

SECONDARY OUTCOMES:
Total Procedure Time | During procedure
Total Radiation Dose | During procedure
Change of LBBAP pacing parameters | From procedure to 1 week
  Threshold @ 0.4ms pulse width, sensing, impedance
Change of LBBAP pacing parameters | From procedure to 1 year
  Threshold @ 0.4ms pulse width, sensing, impedance
Left Ventricular Activation using 2D Speckled Tracking LV Strain (TomTec) | Through study completion, an average of 12 months
LVEF Improvement | From baseline to 12 months
Patient Satisfaction | Through study completion, an average of 12 months
Differences in Quality of Life - EQ5D | From baseline to 12 months
Amount of Tricuspid Regurgitation | Through study completion during echocardiography studies, an average of 12 months
  Measured in mmHg
Change in NTproBNP | From baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No